CLINICAL TRIAL: NCT05163145
Title: Risk Factor for Cholestasis in Neonates receivingTPN At Assiut University Children Hospital
Brief Title: Risk Factor for Cholestasis in Neonates Receiving TPN(Total Parenteral Nutrition)
Acronym: TPN
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mayyada Elsayed Mohamed Hussien (Other)
Responsible Party: Sponsor-Investigator, Mayyada Elsayed Mohamed Hussien, Mayyada Elsayed Mohamed Hussien, Assiut University
Organization: Assiut University (Other)
Other Study IDs: neonates receiveTPN
Record Dates: First submitted 2021-12-06; First posted 2021-12-20 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Neonatal Cholestasis; Total Parenteral Nutrition Effect
Keywords: TPN

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: TPN — early detection of comlications of prolonged TPN on neonatal liver

SUMMARY:
The aim of this study is to evaluate the risk factors of PNAC in neonates

DETAILED DESCRIPTION:
Neonates with prematurity,gastrointestinal dysfunction and very low birth weights are often intolerant to oral feeding.In such infants,the provision of nutrients via parenteral nutrition (PN)becomes necessary for short term survival,as well as long-term health. Wilmore and Dudrick first reported use of parenteral nutrition(PN) for an infant more than 40years ago Soon there after physicians recognized that PN was associated with significant liver changes.In the first reported case of parenteral nutrition-associated conjugated hyperbilirubinemia (PNAC) in a premature infant hepatomegaly was noted on the18thday of fat-free PN and worsened until death on the71st day of life The hyperbilirubinemia manifest in PNAC is thought to occur from impaired hepatic bileflow, an adynamic gallbladder,and an upsurge in release of conjugated bilirubin as an infant matures.Atbirth,preterm neonates havereduced activity of the uridine diphosphate glucuronosyl transferase1A1 liver enzyme(UDPGT)that catalyzes conjugation of bilirubin As the infant develops,UDPGT becomes more functional, increasing hepatocyte efficiency for conjugation.Thus,in combination with cholestasis,and neonatal intestinal absorption of unconjugated bilirubin,more conjugated bilirubin is made available to pass from the liver into circulation. Parenteral nutrition associated cholestasis (PNAC) is the most common form of liver damage in neonates while receiving parenteral nutrition(PN).Its prevalence was reported between10%and 60%in NICU Cholestasisis acommonly described complication of PN. Its etiology is not fully understood and is thought to be multifactorial Proposed mechanisms included altered bile salt metabolisms secondary to prematurity and toxic effect of PN components on the liver the presence or absence of specific components in parenteral nutrition solutions most certainly contributing to the disease mechanism,and gastrointestinal systems .Aggravating factors such as sepsis and duration of bowel rest have also been described

ELIGIBILITY:
Inclusion Criteria:

* Neonates who received PN for ≥14 days

Exclusion Criteria::Neonates with major congenital anomaly, cholestasis at birth,diseases associated with cholestasis (i.e.,inborn errors of metabolism,viral hepatitis,cystic fibrosis and any primary cholestatic liver diseases)that were diagnosed while hospitalized.the possibility of surgical causes of conjugated hyperbilirubinemia(such as biliary atresia,choledochalcyst on abdominal ultrasonography,and hepatobiliary scintigraphy

-

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All neonates who received PN for≥14days and admitted to our children's hospital's NICU
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-03-02 (Estimated)

PRIMARY OUTCOMES:
effect of TPN on neonatal liver | baseline
  TPN associated cholestasis in neonates

IPD SHARING:
Plan to Share IPD: Undecided